## A One-Day ACT Workshop for Emotional Eating Statistical Analysis Plan

Frayn & Knäuper

**September 16, 2018** 

## Statistical Analysis Plan

All analyses will be conducted in SPSS version 24. A repeated measures MANOVA will be conducted to examine the effects of the workshop on the primary outcome (emotional eating) and secondary outcomes (distress tolerance, mindful eating, ACT values application). This analysis will compare changes from baseline to 2-weeks, baseline to 3-months, and 2-weeks to 3-months post-intervention.

Exploratory mediation analyses will be conducted to assess whether or not increases in distress tolerance, mindful eating, and ACT values application mediate the change in emotional eating from baseline to follow-up.

Descriptive statistics will be assessed for the feasibility data (i.e., recruitment, eligibility, attendance, and attrition rates).

Qualitative treatment acceptability data will be subject to thematic analysis as per the procedure outlined by Braun and Clarke (2006).

## References

Braun, V., & Clarke, V. (2006). Using thematic analysis in psychology. *Quantitative*\*Research in Psychology, 3, 77-101